CLINICAL TRIAL: NCT03084497
Title: Effects and Effectiveness of Infant Massage in Motor, Cognitive, Language and Social Developmental in Babies With Syndrome of Down Aged Between 4 and 8 Months
Brief Title: Effects of Infant Massage on Development of Down Syndrome Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Elena Piñero Pinto, PhD, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USeville - EPinto
Record Dates: First submitted 2017-03-08; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Down Syndrome
Keywords: Massage; Development
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving Infant Massage (Experimental): The subjects of this group will receive a total of 5 sessions of Infat Massage.
  Interventions: Procedure: Infant Massage
- Group without intervention (No Intervention): The subjects of this group won´t receive any intervention.

INTERVENTIONS:
Procedure: Infant Massage — The first day, investigators will make the initial assessment of the baby through Psychomotor Development Scale of Early Childhood Brunet- Lézine. Participants will keep the sessions early attention and will participate in the course of Infant Massage, which develop for 5 weeks.
  Infant Massage course will take place with families and is based on the methodology and program of the International Association of Infant Massage ( IAIM ), created by Vimala McClure. The course will consist of 5 sessions (one per week) approximately 90 minutes. Parents will practice everyday the movements learned during the time of the study.
  When the course of Infant Massage finished, Investigators will conduct the final evaluation of the baby, the same way as in the initial evaluation.
  Arms: Group receiving Infant Massage

SUMMARY:
The aim of ths study is to know the effects of infant massage in the maturation of the baby with Down syndrome. Scale Psychomotor Development Early Childhood Brunet-Lézine-Revised will be used to measure the maturational development of the baby with Down syndrome . Investigators will analyze two groups of intervention, the experimental group, in which parents will participate and will apply the knowledge learned in the course of Infant Massage and control, which does not receive the Infant Massage course during the study. Babies in both groups will be evaluated twice, at the beginning of the intervention (pretest) and end it after five weeks (posttest). The study population consists of 32 babies with Down syndrome between 4 and 8 months old.

DETAILED DESCRIPTION:
In this study, the investigators will compare the maturational development of the experimental group Down syndrome babies (will receive infant massage in the period between the two measurements) with the maturational development of the control group Down syndrome babies (will receive infant massage after two measurements). Assess both the development partial motor, cognitive, language and social, and also the maturational development global. Finally, measure also the ratio of development, both in the pretest as on the posttest. The test that will use to measure the development of them babies is the scale of development psychomotor of her first childhood Brunet-Lezine-R. The babies of the study may hay between 4 and 8 months old.

ELIGIBILITY:
Inclusion Criteria:

* Babies with Down Syndrome that received Early Attention.

Exclusion Criteria:

Babies with Down syndrome:

* With associated pathology.
* Adopted.
* Have received infant massage course.

Ages: 4 Months to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change from Developmental Age | At the start of the study (before the first session of Infant Massage and before the asignation of a group) and after the last session of Infant Massage Course (5 weeks)
  Measure by Psychomotor Scale of Developmental in Early Childhood Brunet - Lezine

SECONDARY OUTCOMES:
Change from Developmental coefficient | At the start of the study (before the first session of Infat Massage and before the asignation of the group) and after the last session of Infat Massage Course (5 weeks)
  Measure by Psychomotor Scale of Developmental in Early Childhood Brunet - Lezine

CONTACTS AND LOCATIONS:
Overall Officials: PIÑERO PINTO, Principal Investigator — University of Sevilla
Locations (1):
- University of Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: No